CLINICAL TRIAL: NCT00879697
Title: Effects of Strength Training and Walking Training on Physical Fitness of Patients With Intermittent Claudication
Brief Title: Strength Training in Walking Tolerance in Intermittent Claudication Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Raphael Mendes Ritti Dias, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 44444
Record Dates: First submitted 2009-01-27; First posted 2009-04-10 (Estimated); Results first posted 2009-04-10 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-10

CONDITIONS: Peripheral Arterial Disease; Hypertension; Diabetes
Keywords: peripheral arterial disease; exercise; resistance training; cardiac rehabilitation
MeSH Terms: conditions — Peripheral Arterial Disease; Hypertension; Diabetes Mellitus; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strength training (Active Comparator): Patients who performed strength training. The strength training program was composed by 8 exercises for whole body performed at sub-maximal intensity prescribed according to the patients self-perceived effort
  Interventions: Behavioral: Strength Training
- Walking training (Active Comparator): Patients who performed walking training. The walking training was performed in a treadmill using sub-maximal intensity prescribed based in patients self perceived effort
  Interventions: Behavioral: Walking Training

INTERVENTIONS:
Behavioral: Walking Training — The Walking Training program was performed using a treadmill. In each session, patients performed fifteen 2-min bouts of exercise followed by a 2-min rest interval, as previously described. Walking speed was set in order to induce perceived exertion of 11 to 13 and claudication pain in the last 30 seconds of each exercise bout.
  Other Names: Walk training; Walk exercise
  Arms: Walking training
Behavioral: Strength Training — The strength training program consisted of 8 exercises (leg press, crunches, unilateral knee extension, seated row, unilateral knee flexion, seated bench press, calf raises on leg press, and seated back extension). In each exercise, subjects performed 3 sets of 10 repetitions with a 2-min interval between sets and exercises.
  Other Names: Resistance training; Weight training
  Arms: Strength training

SUMMARY:
Background: Muscle atrophy and reduced leg strength are related to exercise intolerance in patients with intermittent claudication (IC), suggesting that strength training (ST) could improve exercise performance in these patients.

Objective: Analyze the effects of ST in walking capacity in patients with IC comparing with walking training (WT) effects.

Intervention: Patients were randomized into ST and WT. Both groups trained twice a week, for 12 weeks, at the same rate of perceived exertion. ST consisted of 3 sets of 10 repetitions of whole body exercises. WT consisted of 15 two-minute bouts of walking intercalated with 2 minutes of resting.

Measurements: Walking capacity, peak VO2, walking economy, ankle brachial index, ischemic window and knee extension strength

DETAILED DESCRIPTION:
From July 2005 to December 2006, three hundred patients with peripheral arterial disease, who were enrolled in a tertiary center specialized in vascular disease and were able to walk for at least 2 minutes at 2 miles per hour, were invited to a meeting at which explanations about this study were given. 80 patients attended the meeting, 60 of them decided to take part of the study, and 52 attended for the screening tests.

Patients were included in the study if they met the following criteria: Fontaine stage II peripheral arterial disease, symptoms of IC for at least 6 months, ankle/brachial index (ABI) at rest ≤ 0.90 in 1 or 2 legs, reduction of ABI after treadmill test, and exercise tolerance limited by IC. Patients were excluded under the following conditions: presence of chronic lung disease, inability to obtain ABI measurement due to noncompressible vessels, exercise tolerance limited by factors other than claudication (eg, dyspnea or orthopedic problems), poorly controlled blood pressure, presence of electrocardiogram response suggestive of myocardial ischemia during the exercise test, and history of revascularization in the previous year.

Procedures Patients were randomly (by drawing lots) divided into 2 groups: strength (ST, n = 17) and walking (WT, n = 17) training. They were evaluated at baseline (pre-training) and after 12 weeks of exercise training (post-training). During evaluations were assessed exercise tolerance and strength.

Both training programs (ST and WT) were supervised, conducted twice a week, lasted for 12 weeks, and started after a 2-week preconditioning-orientation phase. In both programs, rate of perceived exertion during exercise was kept similar and between 11 to 13 on the15-grade Borg scale. Furthermore, the duration of exercise sessions was prescribed as 30 min of exercise for ST and WT groups.

ELIGIBILITY:
Inclusion Criteria:

* Fontaine stage II peripheral arterial disease(14)
* Symptoms of intermittent claudication for at least 6 months
* Ankle/brachial index (ABI) at rest ≤ 0.90 in 1 or 2 legs
* Reduction of ABI after treadmill test
* Exercise tolerance limited by intermittent claudication

Exclusion Criteria:

* Presence of chronic lung disease
* Inability to obtain ABI measurement due to noncompressible vessels
* Exercise tolerance limited by factors other than claudication (e.g., dyspnea or orthopedic problems)
* Poorly controlled blood pressure
* Presence of electrocardiogram response suggestive of myocardial ischemia during the exercise test
* History of revascularization in the previous year

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-07; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria FN Marucci, PhD, Study Chair — University of Sao Paulo
Locations (1):
- Raphael Dias, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dias RM, Forjaz CL, Cucato GG, Costa LA, Camara LC, Wolosker N, Marucci Mde F. Obesity decreases time to claudication and delays post-exercise hemodynamic recovery in elderly peripheral arterial disease patients. Gerontology. 2009;55(1):21-6. doi: 10.1159/000155219. Epub 2008 Sep 11. PMID 18784409
- [Derived] Grizzo Cucato G, de Moraes Forjaz CL, Kanegusuku H, da Rocha Chehuen M, Riani Costa LA, Wolosker N, Kalil Filho R, de Fatima Nunes Marucci M, Mendes Ritti-Dias R. Effects of walking and strength training on resting and exercise cardiovascular responses in patients with intermittent claudication. Vasa. 2011 Sep;40(5):390-7. doi: 10.1024/0301-1526/a000136. PMID 21948782
- [Derived] Ritti-Dias RM, Wolosker N, de Moraes Forjaz CL, Carvalho CR, Cucato GG, Leao PP, de Fatima Nunes Marucci M. Strength training increases walking tolerance in intermittent claudication patients: randomized trial. J Vasc Surg. 2010 Jan;51(1):89-95. doi: 10.1016/j.jvs.2009.07.118. Epub 2009 Oct 17. PMID 19837534

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2005 to December 2006, three hundred patients with peripheral arterial disease, who were enrolled in a tertiary center specialized in vascular disease and were able to walk for at least 2 minutes (min) at 2 miles per hour (mph), were invited to a meeting at which explanations about this study were given.
Pre-assignment Details: Seven patients did not present symptoms of claudication during the treadmill test, 5 presented electrocardiogram response suggestive of myocardial ischemia, 4 presented exercise tolerance limited by other factors than claudication, and 2 presented poorly controlled blood pressure. All these patients were not included in the study.
Groups:
- Strength Training: Patients who performed strength training. Strength training program consisted of 8 exercises (leg press, crunches, unilateral knee extension, seated row, unilateral knee flexion, seated bench press, calf raises on leg press, and seated back extension). In each exercise, subjects performed 3 sets of 10 repetitions with a 2-minutes interval between sets and exercises.
- Walking Training: Patients who performed walking training. Walking training program was performed using a treadmill. In each session, patients performed fifteen 2-minutes bouts of exercise followed by a 2-minutes rest interval, as previously described. Walking speed was set in order to induce perceived exertion of 11 to 13 and claudication pain in the last 30 seconds (s) of each exercise bout.
Period: Overall Study
Arm/Group | Strength Training | Walking Training
Started | 17 (Seventeen patients achieved inclusion and exclusion criteria) | 17 (Seventeen patients achieved inclusion and exclusion criteria)
Completed | 15 (Two patients did not finish the trial) | 15 (Two patients did not finish the trial)
Not Completed | 2 | 2
Not completed — Physician Decision | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Walking Training: Patients who performed walking training. Walking training program was performed using a treadmill. In each session, patients performed fifteen 2-minutes bouts of exercise followed by a 2-minutes rest interval, as previously described. Walking speed was set in order to induce perceived exertion of 11 to 13 and claudication pain in the last 30 s of each exercise bout.
- Total: Total of all reporting groups
Arm/Group | Strength Training | Walking Training | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (9.5) | 64.6 (8.8) | 65.1 (9.3)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 12 | 10 | 22
Region of Enrollment [Number; unit: participants]
  Brazil | 17 | 17 | 34
Total walking distance [Mean (Standard Deviation); unit: meter] — The maximal walking capacity of patients
  meter | 618 (282) | 572 (231) | 595 (244)

OUTCOME MEASURES:

1. Primary Outcome: Total Walking Distance
Description: The maximal walking distance
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Strength Training | Walking Training
Number analyzed (Participants) | 15 | 15
meter | 618 (282) | 572 (231)
Statistical Analysis 1: Comparison: Strength Training vs Walking Training; The effect of training in both groups were assessed by a 2-way ANOVA (Time x Group) for repeated measures. When significance was obtained, the Newman-Keuls post hoc test was used to identify the differences; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Strength Training | Walking Training
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 2/17 | 2/17
OTHER ADVERSE EVENTS (reported when occurring in more than 3.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strength Training (N=17) | Walking Training (N=17)
Inguinal hernia (Nervous system disorders) | 1 (1) | 0 (0)
Gastrointestinal problems (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diagnose Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diagnose aneurysm (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Our sample was composed of patients with many diseases and taking different medications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No